CLINICAL TRIAL: NCT01795053
Title: Randomized Controlled Trial to Evalualte Effects of Playtraining as Manualized in THOP, a Modulized German ADHD Manual, in 3 to 6 Year Old Children With a Diagnosis of ADHD on ADHD Symptoms and Play Persistence and Intensity
Brief Title: Effects of Playtraining in ADHD Preschoolers on ADHD Symptoms and Play Persistence and Intensity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Manfred Doepfner, university professor, Phd, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: playtrainingADHD
Record Dates: First submitted 2012-08-24; First posted 2013-02-20 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: ADHD
Keywords: ADHD preschoolers; playtraining; child-focused intervention
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- playtraining (Experimental): playtraining is a play based intervention that includes techniques of behavioral management as: structuring of play situation, detailled play planning, definition of behavioral tasks, positive reinforcement, token economy. The intervention is designed to enhance play-persistence and intensity and thereby reduce ADHD symptoms
  Interventions: Behavioral: Experimental: playtraining
- open play session (Placebo Comparator): the open play sessions are conducted in the same rooms, by the same staff and in the same time frame as the experimental sessions. The therapist plays with the child without structuring the sitauation through behavioral tecniques. The play situation is designed to be ineresting and comfortable for the child.
  Interventions: Behavioral: Placebo open play session

INTERVENTIONS:
Behavioral: Experimental: playtraining — playtraining is a play based intervention that includes techniques of behavioral management as: structuring of play situation, detailled play planning, definition of behavioral tasks, positive reinforcement, token economy. The intervention is designed to enhance play-persistence and -intensity and thereby reduce ADHD symptoms
  Arms: playtraining
Behavioral: Placebo open play session
  Arms: open play session

SUMMARY:
A sample of 60 children is randomly assigned to an intervention and a control condition. The intervention group receives 15 sessions of child-focused treatment with play training to enhance play persistence and intensity. The control group receives the same amount of placebo play sessions. The intervention group receives subsequently 15 sessions of parent training. All children are 3 to 6 years old and meet diagnostic criteria for ADD or ADHD. Main hypothesis are a stronger reduction of ADHD symptoms of the child in different settings in the intervention than in the control group. Play-persistence and -intensity should also increase more in the intervention group. An additional effect of a subsequent parent training shall furthermore be tested.

ELIGIBILITY:
Inclusion Criteria: Diagnosis of ADHD or combinde ADHD/ ODD, age 3 to 6, 5 Items regarding play behavior on DSM-IV symptom checklist above 95th percentile, parents motivation to provide 15 to 30 weekly sessions

Exclusion Criteria: Autism Spectrum Disorder, IQ below 80, massive actual impairment, that requests sudden in-patient treatment, school entry in less than 2 months

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2012-02; Primary Completion 2017-07 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
FBB-ADHD-V | 20 minutes
  Symptom checklist, rated by parents and preschool teachers. Standardized quesionnaire based on the DSM-IV diagnostic criteria for ADHD. Specific form for preschoolers with norms from the year 2009

SECONDARY OUTCOMES:
VBV-EL SUBSCALE play productivity and play-intensity | 10 minutes
  questionnaire for preschoolers VBV-EL (=parent version) VBV-ER (=preschool teacher version)focussing items that cover play behavior and restless/ hyperactive behavior

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Doepfner, Prof., PhD, Principal Investigator — University of Cologne
Locations (1):
- University of Cologne, clinic, department for child and adolescent psychtherapy and psychiatry, Cologne, Nordrhein-Westfahlen, Germany